CLINICAL TRIAL: NCT07215936
Title: Dose_dense Capecitabine Schedule [7days on _7days Off] in Colorectal Cancer in Comparison With Standered Regimen
Brief Title: Dose-dense Capecitabine Schedule [7days on _7 Days Off] in Colorectal Cancer in Comparison With Standered Regimen
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aliaa Alaa Abdelrahman, Assisstant lectular of clinical oncology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh_med_25_9___4MD
Record Dates: First submitted 2025-10-04; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Dose_dense capecitabine schedule [7 days on _7 days off ] Compared to standerd regimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A :will receive capecitabine dose dense 1750 mg /m2 7days on treatment and 7 days off (Active Comparator)
  Interventions: Drug: Arm A:Dose_dense Capecitabine in Colorectal cancer
- Arm B will receive capecitabine standard dose 1000mg/m2 2weeks on and 1 week off (Active Comparator)
  Interventions: Drug: Arm B : standard dose Capecitabine

INTERVENTIONS:
Drug: Arm A:Dose_dense Capecitabine in Colorectal cancer — Appling dose _dense Capecitabine 1750mg/m2 for one week then one week off Cycle repeated every 2 weeks
  Arms: Arm A :will receive capecitabine dose dense 1750 mg /m2 7days on treatment and 7 days off
Drug: Arm B : standard dose Capecitabine — Pateints will receive capecitabine 1000 mg/m2 for 2 weeks then one week off
  Arms: Arm B will receive capecitabine standard dose 1000mg/m2 2weeks on and 1 week off

SUMMARY:
Dose_dense Capecitabine Schedule in colorectal cancers

DETAILED DESCRIPTION:
Dose_dense Capecitabine schedule[7 days on_7days off] in colorectal cancer in comparison with standerd regimen

ELIGIBILITY:
Inclusion Criteria:

* patients who diagnosed colorectal cancer Performance status ranging from 0 to 2 Both sexs

Exclusion Criteria:

* pateints with other malignancy Pateints who have other comorbid diseas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
1_Quality of life assessed through EORTC_QLQ_CR29 questionaire | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided